CLINICAL TRIAL: NCT00133783
Title: Intermedin is an Estrogen- Modulated Factor for Reducing Blood Pressure
Brief Title: Pituitary Derived-Intermedin is an Estrogen-Modulated Factor for Reducing Blood Pressure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Other Study IDs: NMRPG34
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2005-10-26 (Estimated); Status verified 2005-05

CONDITIONS: Menopause; Hypertension
Keywords: Intermedin; estradiol; female hypertension; Premenopausal and postmenopausal women; Surgically-induced menopause women; IVF treatment patients
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: intermedin

SUMMARY:
Calcitonin, calcitonin gene-related peptides (CGRPs), adrenomedullin, and amylin belong to a unique group of peptide hormones important for the regulation of calcium balance, neurotransmission, cardiovascular homeostasis, and glucose metabolism. We, the investigators at Chang Gung Memorial Hospital, recently identified intermedin as a novel peptide hormone belonging to this unique peptide ligand family. Adrenomedullin is a 52-amino-acid peptide and is one of the most potent vasodilators. Plasma adrenomedullin is elevated in a variety of pathological conditions such as hypertension, renal failure, heart failure, and septic shock. CGRPα and CGRPβ are 37-amino acid neuropeptides; primarily release from sensory nerves; and play important roles in regulating peripheral vascular tone and controlling blood flow in various organs. Human mature intermedin encodes 40-amino-acid and is expressed mainly in the adrenocorticotrophs of the anterior and intermediate pituitary lobe. Intermedin signals through calcitonin receptor-like receptor (CRLR)/receptor activity-modifying protein (RAMP) receptor complexes, and CRLR/RAMP signaling has been proven to be critical for vascular tone regulation. Based on this finding, we had documented that intraperitoneal administration of intermedin dose-dependently suppressed blood pressure in normal Sprague-Dawley rats. In addition, our preliminary in vitro and in vivo studies demonstrated that ovariectomy lead to a tenfold reduction of intermedin transcript expression in the pituitary in rats whereas subsequent estrogen treatment increased pituitary intermedin expression to a level similar to that of intact rats. Taken together, we propose that pituitary-derived intermedin is regulated by estrogen and exhibits potent hypotensive effects. To address this hypothesis, in Specific Aim 1, we will investigate the regulation of secretion and expression of intermedin in vitro and in vivo using cultured pituitary cells and oophorectomized rats. In Specific Aim 2, we will study the molecular mechanism by which estrogen stimulates intermedin gene expression. In Specific Aim 3, to demonstrate that the estrogen-dependent regulation of intermedin represents a critical link in the regulation of blood pressure in women, we will study the relationship between blood pressure and blood intermedin levels using a cross-sectional study. Our studies will provide a better understanding of the mechanisms by which sex hormones modulate blood pressure and open a new window for postmenopausal hypertension treatment.

DETAILED DESCRIPTION:
Specific Aim:

Validation that intermedin represents an estrogen-regulated vasoactive hormone from the pituitary

Hypothesis:

Intermedin is a mediator of the vaso-regulatory effects of estrogens.

Rationale:

In the Preliminary Study, we showed that intermedin is a pituitary-derived hypotensive factor signaling through CRLR/RAMP receptor complexes in vessel endothelium. Based on studies of related hormones, adrenomedullin and CGRP, intermedin likely reduces blood pressure by exerting a vasodilator effect on vascular beds. Earlier studies have shown that the neuropeptide αCGRP is predominately produced in the sensory neuron, and serotonin can selectively reduce CGRP secretion by activating the endogenous serotonin (type 1 5-HT1) receptor through the calcium signal pathway. Deletion of the CGRP gene in mutant mice (αCGRP-/-) leads to the elevation of mean arterial pressure, heart rate, peripheral vascular resistance and sympathetic nervous activity as compared to wild-type mice. The other related peptide, adrenomedullin (ADM), initially identified from pheochromocytoma, has been shown to be expressed in various tissues including adrenal medulla, cardiovascular tissues, lung, kidney and placenta. Plasma ADM is elevated in various conditions including cardiovascular and renal disorders and septic shock, and it has been hypothesized that ADM may be involved in the control of circulation and body fluid dynamics in various organs. Studies of mice deficient for ADM showed that ADM is indispensable for cardiovascular development. The homozygous knockout ( Adm-/-) mice exhibited an embryonic lethal phenotype.

Earlier studies of the ADM gene promoter have revealed that, in addition to two transcription factors, nuclear factor for interleukin-6 expression (NF-IL6) and activator protein 2 (AP-2), the ADM gene expression is regulated by the hypoxia inducible factor-1 (HIF-1). Under hypoxia conditions, HIF-1 binds to the hypoxia response elements (HRE) in the ADM gene promoter to promote ADM gene expression. Although outside the focus of the present study, we have also detected putative HRE sequences in the intermedin gene promoter and demonstrated that hypoxia conditions stimulate intermedin gene promoter activity, suggesting that HIF-1 could play a role in the regulation of intermedin gene expression. Unlike intermedin, the expression of CGRP and ADM is not actively stimulated by estrogens, suggesting that these two related peptides are not directly associated with the cardiovascular effects of estrogens. In females, 17β-estradiol produced by ovaries is the chief circulating estrogen which increases vasodilatation and inhibits the response of blood vessels to injury. Studies by Mercuro et al. have shown that surgical-induced menopause causes an increase in peripheral vascular resistance and blood pressure. Likewise, a cross sectional study showed that there is a four- fold increase in the incidence of hypertension in postmenopausal women as compared to premenopausal individuals (40% in post menopausal women vs 10% in premenopausal women). The rise in systolic blood pressure per decade was around 5mmHg greater in perimenopausal and postmenopausal women as compared with premenopausal women . In addition to demographic studies, studies have shown that estrogen could dilate coronary and brachial arteries in postmenopausal women. A part of vasodilatation and hypotensive activities of 17β-estradiol could be explained by its ability to modulate the expression of genes known to influence vascular tone and structure, such as ACE, rennin, and angiotension type I (AT1) receptors. However, none of these genes have been shown to be specific direct targets for estrogen receptors and are responsible for the vasoprotective effects of estrogens. Based on our findings that intermedin is a hypotensive factor and contains putative ERE sequence in the promoter region, we propose that intermedin is a pituitary-derived blood pressure modulating factor directly regulated by ovarian estrogens. Based on this understanding, we further hypothesize that the down regulation of intermedin in aging individuals with estrogen deficiency could be responsible for postmenopausal hypertension. Because there is no established animal model suitable for the study of naturally occurring menopause, we will test our hypothesis by studying the relationship between plasma intermedin concentration and blood pressure among women in difference reproductive stages.

Case Selection, Measurement and Analysis of Biophysical and Biochemical Characteristics

Premenopausal and Postmenopausal Group:

Eligible women who visit OB/GYN physicians will be invited for an interview. They will be questioned about general characteristics, lifestyle habits (smoking, alcohol consumption, physical activity), and medical history. During the interview, blood pressure will be measured three times on the right arm, while the participant is seated. A woman is considered as post menopausal if her menses have naturally ceased for 12 months (or more), or if she has bilateral oophorectomy or hysterectomy without bilateral oophorectomy and aged more than 55 years. Office BP will be measured using a mercury sphygmomanometer according to the recommendations of the American Society of Hypertension (average the three BP readings after 5 min of quiet sitting position). Biophysical and biochemical characteristics will be measured including the last menses period, age, BMI, serum glucose (AC and PC), serum and urine creatinine, plasma total cholesterol, HDL, LDL, triglycerides, FSH, LH, 17β-estradiol, progesterone, TSH, intermedin, and prolactin. Blood specimens from individual subjects will be analyzed in a single assay to minimize variations. Odds ratios (ORs) of elevated blood pressure and the corresponding 95% confidence intervals (CIs) will be computed after allowance for age. Furthermore, in order to take into account potential reciprocal confounding effects of variables considered, factors significantly related with elevated blood pressure risk in the age adjusted analysis will be subsequently included in multiple logistic regression models fitted by the method of maximum likelihood. Women asking for annually regular pap smear examinations without any medical disease will be eligible for this study group.

The reproductive stages will be assigned as:

* Premenopausal: no reported change in menstrual cycle pattern;
* Early peri-menopausal: reported change in menstrual cycle frequency in preceding year with a bleed in the preceding 3 months;
* Late peri-menopausal: no menses in the preceding 3-11 months;
* Postmenopausal: no menses in the preceding 12 months.

Surgically-Induced Menopausal Group:

This protocol will include fertile women who suffer from ovarian pathology without other medical disease and are scheduled to undergo bilateral oophorectomy associated with or without hysterectomy. Patients who suffer from uterine pathology and undergo hysterectomy only will serve as controls. Blood pressure and all biochemical characteristics will be measured one week before surgery and 1, 3, 6 and 12 months after operation. All individual measurements will be blinded as to the hysterectomized/oophorectomized status of the patients. The entire data group will be reported as mean ± SE. Differences in vascular parameters between oophorectomized women and controls and between values recorded prior to and following surgery will be assessed using paired and unpaired Student's t-tests.

ART Group:

Women in ART treatment due to male or tubal factor will be included. The day 3 hormone level (E2, progesterone, FSH, LH, TSH, prolactin, inhibin A, inhibin B and activin) and blood pressure will be measured one month before ART treatment. After gonadotropin administration, all the hormone and blood pressure changes will be measured and recorded at day 3, day 7 and the day before hCG injection as well as the day of oocyte retrieval. All biophysical and biochemical characteristics will continue to follow up on the 15th day after embryo transfer and to the end of the first trimester in the pregnancy group.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women: no reported change in menstrual cycle pattern
* Early peri-menopausal women: reported change in menstrual cycle frequency in preceding year with a bleed in the preceding 3 months
* Late peri-menopausal women: no menses in the preceding 3-11 months
* Postmenopausal women: no menses in the preceding 12 months
* Patients who received oophorectomy
* Patients who received hysterectomy for benign uterus tumor
* Patients underwent assisted reproductive technology (ART).

Exclusion Criteria:

* Patients underwent chemotherapy or radiotherapy in past two years

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2005-05; Study Completion 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Chialin Chang, M.D., Principal Investigator — Chang Gung Memorial Hospital, Department of OB/GYN, 5. Fu-Hsing St. Kwei-Shan, Tao-Yuan, Taiwan, ROC
Locations (1):
- Chailin Chang, Kwei-Shan, Tao-Yuan, Taiwan

REFERENCES:
- [Background] Lin Chang C, Roh J, Park JI, Klein C, Cushman N, Haberberger RV, Hsu SY. Intermedin functions as a pituitary paracrine factor regulating prolactin release. Mol Endocrinol. 2005 Nov;19(11):2824-38. doi: 10.1210/me.2004-0191. Epub 2005 Jul 7. PMID 16002435